CLINICAL TRIAL: NCT00632567
Title: Anal Incontinence After Delivery. Secondary Prevention With Caesarean Section.
Brief Title: EPIC :Anal Incontinence After Delivery. Secondary Prevention With Caesarean Section.
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P060246
Record Dates: First submitted 2008-02-28; First posted 2008-03-10 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Fecal Incontinence
Keywords: Anal incontinence; First delivery was traumatic; No anal incontinence
MeSH Terms: conditions — Fecal Incontinence; Encopresis | interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): caesarean section
  Interventions: Procedure: caesarean section
- 2 (Active Comparator): vaginal delivery
  Interventions: Procedure: vaginal delivery

INTERVENTIONS:
Procedure: caesarean section — caesarean section for second delivery if the first had to be traumatic after forceps with anal sphincter rupture diagnosed with anal endosonography.
  Arms: 1
Procedure: vaginal delivery — vaginal delivery for second delivery if the first had to be traumatic after forceps with anal sphincter rupture diagnosed with anal endosonography.
  Arms: 2

SUMMARY:
Anal incontinence is frequent and treatment is difficult. One of the most important reasons is traumatic delivery. 10 % of women develop anal incontinence after first delivery. This incidence is higher after second vaginal delivery, particularly if the first delivery caused break in the anal sphincter. One possibility to avoid anal incontinence is the caesarean section. So, do the investigators have to recommend caesarean section for second delivery if the first was traumatic? But caesarean section had a morbidity. Actually, the choice between the delivery modalities is very subjective.

DETAILED DESCRIPTION:
Anal incontinence is frequent and treatment is difficult. One of the most important reasons is traumatic delivery. 10 % of women develop anal incontinence after first delivery. This incidence is higher after second vaginal delivery, particularly if the first delivery caused break in the anal sphincter. One possibility to avoid anal incontinence is the caesarean section.

So, do the investigators have to recommend caesarean section for second delivery if the first was traumatic? But caesarean section had a morbidity. Actually, the choice between the delivery modalities is very subjective. It seems to be very useful to compare, in randomized controlled study, global morbidity of caesarean section and vaginal delivery for second delivery if the first had to be traumatic after forceps with anal sphincter rupture diagnosed with anal endosonography. In start of study, all women were included, for randomisation ("section cesarean prophylactic" versus "vaginal delivery") if an anal sphincter rupture is diagnosed with anal endosonography before second delivery. . Currently, in case of refusal randomisation, women are proposed to participate to the ancillary study (cohort study).

The primary endpoint is comparison of median incontinence score of VAISEY in the two arms after 6 months. The secondary endpoints are urinary incontinence, quality of life and global morbidity between the two arms after second delivery. The investigators estimated, needing 123 women in each arm.

Hospital investigators are: BICHAT Claude Bernard (Pr LUTON), Armand Trousseau (Pr BENIFLA), Jean VERDIER (Pr CARBILLON), BEAUJON (Pr LUTON), Louis MOURIER (Pr MANDELBROT), Versailles (Dr PANEL). Inclusion will be for 6 years and 9 months. Women will be included during the last trimester and evaluation will be perform on 8 weeks, 6 and 12 month after delivery.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Having health insurance
* Second pregnancy
* Inclusion in the third trimester
* First delivery was traumatic
* No anal incontinence
* Accept to participate, sign the informed consent
* Prior medical examination

Exclusion Criteria:

* Monitoring impossible
* Woman who have an anal operation
* Caesarean section
* First delivery with anal break stage 4
* Indication of a scheduled caesarean section not for proctologic reason
* Patient physically, mentally or legally incompetent to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2008-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is comparison of median incontinence score of VAIZEY in the two arms after 6 months. | 6 months

SECONDARY OUTCOMES:
Incontinence scores in the two arms after 6/8 weeks and 6 month, transitional anal incontinence after delivery urinary incontinence 6 and 12 month after the delivery, sexual score(IFSI)global morbidity between the two arms after anal endoscopy | 6 month and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Laurent ABRAMOWITZ, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital BICHAT, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided